CLINICAL TRIAL: NCT06374758
Title: ACCELERATE a Multisite Prospective Hybrid (Effectiveness-implementation) Type 2 Design, Single-arm, Mixed-methods Study of a Simplified Accelerated ART Initiation Protocol for People With HIV Who Are Out of Care.
Brief Title: Accelerated ART Initiation for PWHIV Who Are Out of Care
Acronym: ACCELERATE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Dima Dandachi, Assistant Professor, Medical Director of HIV treatment and prevention, Columbia/Boone County Health and Human Services, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MU-2096449
Record Dates: First submitted 2024-03-27; First posted 2024-04-19 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections; ART; Noncompliance, Patient
MeSH Terms: conditions — HIV Infections; Patient Compliance | interventions — bictegravir; Emtricitabine; tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Accelerate Model of Care (Experimental): Contact is established by the study team
  The patient is provided with a telehealth appointment with an HIV care provider within 24 business hours of contact
  At the time of enrollment/initial clinic visit, patients who meet the inclusion and exclusion criteria will be enrolled in the study
  The HIV care provider will prescribe B/F/TAF to their pharmacy of choice.
  B/F/TAF is dispensed by the designated study pharmacist and mailed to the patient as a free 30-day starter pack to allow time for benefits verification.
  A telephone follow-up call by the study team will be conducted within 2 - 4 weeks from the initial clinical visit to assess any adverse events, tolerability, and adherence.
  Hand-off to HIV clinic to establish care within 4 weeks. Lab results will be drawn during clinic per HIV care provider which might include CBC, CMP, HIV-1 RNA, CD4, and genotype resistance testing when clinically indicated by the HIV care provider.
  Interventions: Other: The Accelerate model of care; Drug: bictegravir/emtricitabine/tenofovir alafenamide 50/200/25 mg

INTERVENTIONS:
Other: The Accelerate model of care — Contact is established by the study team
  The patient is provided with a telehealth appointment with an HIV care provider within 24 business hours of contact
  At the time of enrollment/initial clinic visit, patients who meet the inclusion and exclusion criteria will be enrolled in the study
  The HIV care provider will prescribe B/F/TAF to their pharmacy of choice.
  B/F/TAF is dispensed by the designated study pharmacist and mailed to the patient as a free 30-day starter pack to allow time for benefits verification.
  A telephone follow-up call by the study team will be conducted within 2 - 4 weeks from the initial clinical visit to assess any adverse events, tolerability, and adherence.
  Hand-off to HIV clinic to establish care within 4 weeks. Lab results will be drawn during clinic per HIV care provider which might include CBC, CMP, HIV-1 RNA, CD4, and genotype resistance testing when clinically indicated by the HIV care provider.
Drug: bictegravir/emtricitabine/tenofovir alafenamide 50/200/25 mg — Same as above, it is the same intervetion

SUMMARY:
The main purpose of the study is to evaluate the effectiveness, of the ACCELERATE model of care to achieve HIV viral suppression at Week 24. The study will also assess the acceptability, appropriateness, feasibility, and sustainability of the ACCELERATE model of care. The ACCELERATE model combines a standardized method for outreach, the use of telehealth for rapid access to an HIV care provider, a simplified pre-approved HIV regimen, a free 30-day medication starter supply, and re-linkage to medical care.

DETAILED DESCRIPTION:
This is a multisite prospective hybrid (effectiveness-implementation) type 2 design, single-arm, mixed-methods study of a simplified accelerated ART initiation protocol for People with HIV who are out of care.

The investigators will assess the effectiveness of achieving HIV viral suppression defined as HIV RNA < 200 copies/mL at week 24 with B/F/TAF (Biktarvy) as a rapid start for PWH who are out of care.

The investigators will also study the acceptability, feasibility, and sustainability of an innovative model of care that combines a standardized method for outreach, the use of telehealth for rapid access to an HIV care provider, a simplified pre-approved ART regimen, a mailed free starter, and re-linkage to care As an implementation science study, the investigators will explore the methods and factors influencing the successful integration of evidence-based practices across diverse settings.

This study will also ask the staff implementing the ACCELERATE approach about its ease of use, feasibility, compliance, and possible obstacles to its application.

ELIGIBILITY:
PLWH Inclusion criteria: Participants must meet ALL the following inclusion criteria

1. 18 years or older at the time of obtaining the informed consent
2. Speaks English
3. Able to give consent which includes the ability to understand and comply with study requirements and instructions as judged by clinic or study staff
4. HIV-1 infection as documented by positive HIV test (positive laboratory HIV 1/2 Antibody differentiation assay or detectable HIV -1 RNA)
5. Out of care, defined as not had a medical visit with an HIV care provider with prescribing privileges for ≥6 months AND not receiving ART for ≥1 month (by self-report)

Site Staff Inclusion criteria:

Participants must meet ALL the following inclusion criteria

1. 18 years or older at the time of obtaining the informed consent
2. HIV care providers, case managers, pharmacists, or administrators involved in administrative or clinical aspects of the intervention at participating sites
3. Understand the long-term commitment to the study and be willing to participate
4. Have adequate resources to complete assessments for the duration of the study

Exclusion criteria PLWH Exclusion criteria: Participants who meet ANY of the following criteria are excluded

1. Biktarvy (B/F/TAF) contraindicated or not recommended

   1. Known history of chronic kidney disease (creatinine clearance <30 mL/min) using Cockcroft-Gault formula AND not on chronic dialysis
   2. Known history of allergy to B/F/TAF components
   3. Known history of intermediate-high level resistance to B/F/TAF components (score ≥30 on Stanford HIV Drug Resistance Algorithm) in the available medical record (not having a prior genotype or having M184V/I mutation is NOT an exclusion criterion)
   4. Concomitant use of contraindicated medications: using drug interaction database either Lexicomp® Drug Interactions (category X Avoid combination) or Liverpool HIV Interactions Checker (category Do not Co-administer) or study drug label (USPI) as reference for list of contraindicated meds.
   5. Pregnant (by self-report) or planning to become pregnant while enrolled in the study
2. HIV-2 infection
3. PLWH who are breastfeeding and are not on ART or taking ART without virologic suppression since breastfeeding will not be recommended.
4. Active opportunistic infections that would require a delay of ART as judged by the HIV care provider and based on current Guidelines for the Prevention and Treatment of Opportunistic Infections in Adults and Adolescents with HIV: such as cryptococcal and Tuberculous meningitis, and CMV retinitis.16
5. Not residing in the state of Missouri at the time of the study or planning to relocate during the study period
6. Incarcerated at the time of the study enrollment.

Site Staff Exclusion criteria:

1) Moving practice location or job relocation within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of the ACCELERATE model of care to achieve HIV viral suppression at Week 24. | 24 weeks
  Proportion of participants who have plasma HIV RNA <200 c/mL at Week 24 (observed analysis)
To study the change over time in the acceptability of the ACCELERATE model of care in patient and staff participants. | 1 year
  Quantitative Change in the mean scores of the Acceptability of Intervention Measure (AIM) scores at Weeks 24, and 48 by PLWH Change in the mean scores of the Acceptability of Intervention Measure (AIM)scores from baseline at Week 48 by Staff participants.
  Min score: 4 (worst) Max score: 20 (best)
To study the change over time in appropriateness of the ACCELERATE model of care in patient and staff participants | 1 year
  Quantitative Change in the mean scores of the Intervention Appropriateness Measure (IAM) scores at Weeks 24, and 48 by PLWH Change in the mean scores of the Intervention Appropriateness Measure (IAM) scores from baseline at Week 48 by Staff participants.
  Min score: 4 (worst) Max score: 20 (best)
To study the change over time in feasibility of the ACCELERATE model of care in staff participants | 1 year
  Quantitative Change in the mean scores of the Feasibility of Intervention Measure (FIM) scores from baseline at Weeks 24, and 48 by PLWH Change in the mean scores of the Feasibility of Intervention Measure (FIM) scores from baseline at Week 48 by Staff participants.
  Min score: 4 (worst) Max score: 20 (best)
To study the change over time in sustainability of the ACCELERATE model of care in staff participants | 1 year
  Quantitative Mean overall score of Clinical Sustainability Assessment Tool (CSAT) and change from baseline at Week 48 by Staff participants.
  Min score: 0 (worst) Max score: 147 (best)
Qualitative data | 1 year
  One-on-one Semi-structured interviews with PLWH and Staff Participants at end of study.

SECONDARY OUTCOMES:
To evaluate the effectiveness of the intervention to achieve HIV viral suppression at week 48 using ACCELERATE model of care. | 1 year
  The proportion of participants who
  * Have HIV RNA <50 c/mL at Week 24 and 48 (observed analysis)
  * Have HIV RNA <50 c/mL at Week 24 and 48 using Intent-to-treat (ITT) analysis, including all participants who have received at least one dose of B/F/TAF.
To assess change in patient experience (PROs) and satisfaction for participants using the ACCELERATE model of care | 1 year
  Change from baseline in overall Consumer Assessment of Healthcare Providers and Systems-Clinician and Group (CAHPS®-CG)19 at Weeks 24, and 48.
  The CG-CAHPS Adult Visit Survey contains 42 items, of which 13 are used to create three composites which assess Access to Care (five items), Doctor Communication (six items), and Courteous/Helpful Staff (two items). The survey also includes two questions that ask respondents (1) to rate their doctor, and (2) report if they would recommend the doctor's office to family and friends. In addition, respondents are asked about their overall health, age, gender, and education.
  Source: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3480671/
To assess change in health-related quality of life (HRQoL) | 1 year
  Change from baseline in Physical Component Summary (PCS) score and & Mental Component Summary (MCS) of the Short Form (SF-36®)20 at Weeks 24, and 48.
  Min score: 0 (worst) Max score: 3600 (best) source: https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/scoring.html
To measure the change in patients' satisfaction with the HIV treatment regimen B/F/TAF | 1 year
  Change from week 4 in the overall score of the treatment Satisfaction Questionnaire21 at Weeks 24, and 48. To account for a potential ceiling effect that may occur due to the baseline, the appropriate version of the HIV treatment satisfaction questionnaire (HIVTSQ) (status or change) will be used.
  Min score: 0 (worst) Max score: 60 (best)
To measure Retention in Care | 1 year
  * The proportion of participants who completed their Week 24 and Week 48 visit
  * The proportion of participants who met the definition of the Health Resources & Services Administration (HRSA) HIV/AIDS Bureau Annual RIC22 at Week 48 (had at least 2 encounters within the 12-month measurement year).
To assess the adherence to the study treatment | 1 year
  Using the 3-item self-reported adherence measure Weeks 4, 24, and 48.
  The 3 items are:
  1. Number of days of missed treatment
  2. In the last 30 days, how good a job did you do at taking your HIV medicines in the way that you were supposed to?
  3. In the last 30 days how often did you take your HIV medicines in the way that you were supposed to?
  For analyses item responses for the three adherence items will be linearly transformed to a 0-100 scale with zero being the worst adherence, and 100 the best. Therefore:
  Min score: 0 (worst) Max score: 300 (best) source: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5071118/
To study the virologic response of using B/F/TAF as first line regimen in ACCELERATE model of care. | 1 year
  Incidence of treatment-emergent genotypic resistance to B/F/TAF or any other ART, in participants meeting confirmed virologic failure (inability to achieve HIV RNA <200 c/mL at week 24 or to maintain HIV RNA <200 c/mL after virologic suppression).
To study the immunologic response of using B/F/TAF as first line regimen in ACCELERATE model of care. | 1 year
  Change from baseline/week 4 in CD4 cell counts at Weeks 24 and 48.
To assess staff impact of ACCELERATE model of care on staff satisfaction | 1 year
  Using the staff questionnaire at baseline and week 48 min score: 5 (worst) max score: 25 (best)
To assess staff impact of ACCELERATE model of care on staff burnout | 1 year
  Using the staff questionnaire at baseline and week 48 Min score: 10 (best) Max score: 70 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Dima Dandachi, MD, MPH, Principal Investigator — University of Missouri-Columbia
Locations (4):
- United States (4):
  - University of Missouri-Columbia, Columbia, Missouri
  - KC Care Health Center, Kansas City, Missouri
  - AIDS Project of the Ozarks, Springfield, Missouri
  - NOVUS Health, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No
Unauthorized disclosure of personal information could lead to damage to the subjects' reputation. Subjects may experience embarrassment and social stigmatization if private details about their health conditions, behaviors, or personal history become known to others in their community or social circles. The loss of privacy may lead to psychological distress, anxiety, or emotional harm, can expose individuals to discrimination or prejudice. Fear of privacy breaches may result in reduced willingness of individuals to participate in future research studies, impacting the scientific community's ability to conduct meaningful research.
  To mitigate these risks, we incorporated robust privacy protection measures, including secure data storage and de-identification of data.